CLINICAL TRIAL: NCT05144984
Title: Investigation of the Safety and Efficacy of Semaglutide s.c. in Combination With NNC0480-0389 in Participants With Type 2 Diabetes - a Dose Finding Study
Brief Title: A Research Study Looking at How Well a Combination of the Medicines Semaglutide and NNC0480-0389 Works in People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9389-4606; U1111-1259-2741 (Other: World Health Organization (WHO)); 2020-004863-14 (EudraCT Number); jRCT2031210474 (Other: Japanese Registration Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 2.4 mg semaglutide + 2.4 mg NNC0480-0389 (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. semaglutide.
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- Placebo (semaglutide) + placebo ( 2.4 mg NNC0480-0389) (Placebo Comparator): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of placebo (NNC0480-0389) co-administered with s.c. placebo (semaglutide).
  Interventions: Drug: Placebo (NNC080-0389); Drug: Placebo (semaglutide)
- 2.4 mg semaglutide + 7.2 mg NNC0480-0389 (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. semaglutide
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- 2.4 mg semaglutide + 12.0 mg NNC0480-0389 (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. semaglutide
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- 2.4 mg semaglutide + 21.6 mg NNC0480-0389 (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. semaglutide
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- NNC0480-0389 + placebo (semaglutide) (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. placebo (semaglutide)
  Interventions: Drug: NNC0480-0389; Drug: Placebo (semaglutide)
- Placebo (semaglutide) + placebo ( 7.2 mg NNC0480-0389) (Placebo Comparator): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of placebo (NNC0480-0389) co-administered with s.c. placebo (semaglutide).
  Interventions: Drug: Placebo (NNC080-0389); Drug: Placebo (semaglutide)
- Placebo (semaglutide) + placebo ( 12.0 mg NNC0480-0389) (Placebo Comparator): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of placebo (NNC0480-0389) co-administered with s.c. placebo (semaglutide).
  Interventions: Drug: Placebo (NNC080-0389); Drug: Placebo (semaglutide)
- Placebo (semaglutide) + placebo ( 21.6 mg NNC0480-0389) (Placebo Comparator): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of placebo (NNC0480-0389) co-administered with s.c. placebo (semaglutide).
  Interventions: Drug: Placebo (NNC080-0389); Drug: Placebo (semaglutide)
- Semaglutide 2.4 mg + placebo (NNC0480-0389) (Experimental): subjects will receive once weekly subcutaneous (s.c., under the skin) dose of placebo (NNC0480-0389) co-administered with s.c. semaglutide.
  Interventions: Drug: Semaglutide; Drug: Placebo (NNC080-0389)

INTERVENTIONS:
Drug: NNC0480-0389 — A weekly dose of NNC0480-0389, dose increased in each cohort. The study will last for about 41weeks.
  Arms: 2.4 mg semaglutide + 12.0 mg NNC0480-0389; 2.4 mg semaglutide + 2.4 mg NNC0480-0389; 2.4 mg semaglutide + 21.6 mg NNC0480-0389; 2.4 mg semaglutide + 7.2 mg NNC0480-0389; NNC0480-0389 + placebo (semaglutide)
Drug: Semaglutide — A weekly dose of semaglutide, same dose in each cohort. The study will last for about 41weeks.
  Arms: 2.4 mg semaglutide + 12.0 mg NNC0480-0389; 2.4 mg semaglutide + 2.4 mg NNC0480-0389; 2.4 mg semaglutide + 21.6 mg NNC0480-0389; 2.4 mg semaglutide + 7.2 mg NNC0480-0389; Semaglutide 2.4 mg + placebo (NNC0480-0389)
Drug: Placebo (NNC080-0389) — A weekly dose of placebo (NNC0480-0389). The study will last for about 41weeks.
  Arms: Placebo (semaglutide) + placebo ( 12.0 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 2.4 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 21.6 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 7.2 mg NNC0480-0389); Semaglutide 2.4 mg + placebo (NNC0480-0389)
Drug: Placebo (semaglutide) — A weekly dose of placebo (semaglutide). The study will last for about 41weeks.
  Arms: NNC0480-0389 + placebo (semaglutide); Placebo (semaglutide) + placebo ( 12.0 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 2.4 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 21.6 mg NNC0480-0389); Placebo (semaglutide) + placebo ( 7.2 mg NNC0480-0389)

SUMMARY:
This study is looking at semaglutide in combination with a potential new medicine (NNC0480-0389) in people with type 2 diabetes.

The study is being conducted to see how well semaglutide, in combination with different doses of NNC0480-0389, work to lower blood sugar levels. Results from this study will be used to select the doses of the two medicines for other studies.

Participants will either get:

Semaglutide (a medicine doctors can already prescribe for treatment of type 2 diabetes) in combination with NNC0480-0389 (a potential new medicine) or placebo (a 'dummy' medicine that looks like the medicines but without any medicine).

NNC0480-0389 alone, or semaglutide alone which treatment participant get is decided by chance.

Participant will need to take 2-3 injections once every week during the study. One injection will be with semaglutide or placebo and 1-2 injections will be with NNC0480-0389 or placebo.

Participant must inject the study medicines themself into the stomach, thigh, or upper arm.

The study will last for about 41weeks. Participant will have 20 clinic visits. Participant will have blood samples taken at all clinic visits. At 3 clinic visits, participant will also have an electrocardiogram (ECG). This is a test to check participants heart. Participant will have their eyes checked before or at the start of the study and at the end of the study.

Women can only take part in the study if they are not able to become pregnant

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days before screening
* Participants treated with diet and exercise as monotherapy or in combination with stable daily dose(s) greater than or equal to 90 days before screening of any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose
* HbA1c 7.0-10.0% (53-86 mmol/mol) (both inclusive)
* BMI greater than or equal to 25 and below 40 kg/m^2

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 days and prior insulin treatment for gestational diabetes are allowed
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic cardiovascular, gastrointestinal, or endocrinological conditions (except conditions associated with T2D)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to visit 24 (week 34)
  percentage-point

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG) | From baseline (week 0) to visit 24 (week 34)
  measured in mmol/L
Change in body weight (kg) | From baseline (week 0) to visit 24 (week 34)
  measured in kg
Change in body weight (%) | From baseline (week 0) to visit 24 (week 34)
  measured in percent
Change in waist circumference | From baseline (week 0) to visit 24 (week 34)
  measured in cm
Change in systolic blood pressure (SBP) | From baseline (week 0) to visit 24 (week 34)
  measured in mmHg
Relative change in total cholesterol | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in very-low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in triglycerides | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in free fatty acids | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in Apolipoprotein B (ApoB) | From baseline (week 0) to visit 24 (week 34)
  ratio
Relative change in high sensitivity C-Reactive Protein (hsCRP) | From baseline (week 0) to visit 24 (week 34)
  ratio
Number of treatment-emergent adverse events (TEAEs) | From baseline (week 0) to visit 25 (week 39)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (129):
- United States (71):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Synexus Clinical Research, Glendale, Arizona
  - University of Arizona/Banner Health, Phoenix, Arizona
  - American Clinical Trials, Buena Park, California
  - San Fernando Valley Hlth Inst, LLC, Canoga Park, California
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - Headlands Research California, LLC, Escondido, California
  - Valley Research, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Velocity Clinical Research San Diego, La Mesa, California
  - First Valley Med Grp Lancaster, Lancaster, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Artemis Insitute for Clin Res, Riverside, California
  - Artemis Institute for Clin Res, San Diego, California
  - Shahram Jacobs MD Inc., Sherman Oaks, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Northeast Research Institute, Jacksonville, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - South Broward Research LLC, Miramar, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Headlands Research - Sarasota, Sarasota, Florida
  - Appalachian Clinical Res LLC, Adairsville, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Macoupin Research Group, Gillespie, Illinois
  - UnityPoint Health-Diabetes Care Center, Peoria, Illinois
  - Clin Invest Spec, Inc, Wauconda, Illinois
  - Iowa Diabetes & Endo Res Ctr, West Des Moines, Iowa
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Centex Studies, Inc._Lake Charles, Lake Charles, Louisiana
  - Endo And Metab Cons, Rockville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - Princeton Endo Assoc, Princeton, New Jersey
  - Premier Research Inc., Trenton, New Jersey
  - AMC Community Endocrinology, Albany, New York
  - Mid Hudson Med Res-New Windsor, New Windsor, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Albert J Weisbrot, Mason, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Intend Research, Norman, Oklahoma
  - Essential Medical Research LLC, Tulsa, Oklahoma
  - CCT Research, Hatboro, Pennsylvania
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Centex Studies, Inc., Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Centex Studies, Houston, Texas
  - Quality Research Inc, San Antonio, Texas
  - VIP Trials_San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Advanced Research Institute, Ogden, Utah
  - York Clinical Research LLC, Norfolk, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Bulgaria (7):
  - Medical centre Zdrave 1 OOD, Kozloduy
  - IPMC - Dr. Elizabeta Dimitrova, Petrich
  - UMHAT Aleksandrovska, Sofia
  - Medical centre - Doverie AD, Sofia
  - UMHAT Sofiamed EAD, Sofia
  - Prevencia - 2000 - MCOC OOD, Stara Zagora
  - Medical center Berbatov, Yambol
- Denmark (3):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Center for Klinisk Metabolisk Forskning, Hellerup
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
- Greece (8):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - Iatriko Psychicou Private Clinic, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
- Hungary (13):
  - PTE-AOK II. Belgyogyaszati Klinika es Nephrologiai Centrum, Pécs, Baranya Vármegye
  - Debreceni Egyetem Belgyógyászati Klinika, Debrecen, Hajdú-Bihar
  - Békés Megyei Központi Kórház - dr. Réthy Pál Tagkórház, Békéscsaba
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - SOTE ÁOK I. sz. Belgyógyászati és Onkológiai Klinika, Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MED-TIMA Kft., Budapest
  - MH Egészségügyi Központ, Budapest
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika D épület, Debrecen
  - Békés Megyei Központi Kórház, Gyula
  - Kaposi Mór Oktató Kórház, Kaposvár
  - Vas Vármegyei Markusovszky Egyetemi Oktatókórház, Szombathely
  - Szent Borbála Kórház, Tatabánya
- Japan (6):
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Yoshimura clinic, Kumamoto
  - Kansai Electric Power Hospital_Center for Diabetes, Osaka
  - Tokyo Center Clinic, Tokyo
  - ToCROM Clinic, Tokyo
  - Higashi-shinjuku clinic, Tokyo
- Poland (13):
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Globe Badania Kliniczne Sp. z o.o., Kłodzko
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - FutureMeds Sp. z o.o. Lodz, Lodz
  - Diabetica Sp. z o.o., Nysa
  - Centrum Medyczne dr Sudnik, Sokółka
  - Osrodek Badan Klinicznych Clinsante, Torun
  - Centrum Medyczne AMED Warszawa, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - FutureMeds Sp. z o.o., Wroclaw
  - SPSK nr 1 im. prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, ul. 3-go Maja 13/15 41-800 Zabrze, Zabrze
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Russia (4):
  - Tumen State Medical University, Tyumen, Russia
  - LLC RC Medical, Novosibirsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Medinet LLC, Saint Petersburg
- Serbia (4):
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocr, Kragujevac

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com